CLINICAL TRIAL: NCT05051774
Title: The Effectiveness of a Motivated, Action-based Intervention on Improving Physical Activity Level, Exercise Self-efficacy and Cardiovascular Risk Factors of Coronary Heart Disease Patients: A Randomized Controlled Trial
Brief Title: Effectiveness of a Motivated, Action-based Intervention on Health Outcomes of Coronary Heart Disease Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study had been suspended last year due to COVID-19 pandemic.
Sponsor: Karthikesu Karthijekan (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Karthikesu Karthijekan, Principal Investigator, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CREC Ref.No.:2020.678 -T
Record Dates: First submitted 2021-09-01; First posted 2021-09-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; Physical activity level; Exercise self-efficacy
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: A single-blind parallel randomized control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcomes assessors only will be blinded in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to usual care, the intervention group will receive the 12 weeks intervention consists of three monthly group education and center-based group exercise followed by 20 minutes of individualized telephone follow-up at weeks 3, 7, and 11.
  Interventions: Behavioral: 1. Education; Behavioral: 2. Exercise; Behavioral: 3. Telephone follow-up
- Control Group (No Intervention): The control group will receive the usual care provided in the study hospital included an unstructured health education conducted by a nurse on healthy lifestyle and health assessment and brief unstructured health education on their conditions, focusing on the risk factors management and stress management by the cardiologist.

INTERVENTIONS:
Behavioral: 1. Education — Three monthly face-to-face group education with 8 to10 participants using a validated educational booklet will be provided by the researcher at the study hospital.
  Arms: Intervention Group
Behavioral: 2. Exercise — The exercise intervention comprised of two elements as follows:
  1. Three monthly hospital-based supervised group exercise consists of 8 to 10 participants. First two sessions: warm-up exercise-5 minutes, brisk walking-20 minutes at low intensity with music, and cool-down exercise-5 minutes. Third session: brisk walking for 30 minutes at moderate intensity with music.
  2. Twelve-weeks home-based exercise: The participants will be asked to continue the exercise performed in the previous week at the hospital with music at least five times per week.
  Arms: Intervention Group
Behavioral: 3. Telephone follow-up — A 20-minutes telephone follow-up at weeks 3, 7, and 11 for strengthening the volition of the participant to perform the exercise and follow the healthy diet at home.
  Arms: Intervention Group

SUMMARY:
Coronary heart disease (CHD), the major group of cardiovascular disorders, is the leading cause of cardiac-associated mortality, causing >9 million death in 2016. American Heart Association (AHA) and the American College of Cardiology Foundation (ACCF) recognized that lifestyle modification including physical activity is the class one-level recommendation for secondary prevention and risk reduction therapy for patients with CHD. The assessment of physical activity and confidence in performing exercise for patients with CHD will help healthcare professionals to develop and implement the appropriate intervention to enhance patients' confidence in performing exercise and physical activity to promote and maintain their health.

With the increasing morbidity and mortality from CHD, especially in low and middle-income countries, secondary prevention including exercise-based cardiac rehabilitation (CR) plays an important role to improve the prognosis of CHD patients. High prevalence of physical inactivity, unhealthy dietary practices, poor control of blood glucose, blood pressure (BP), blood lipid, and body weight (BW) was found among CHD patients in the world as well as in Sri Lanka. Therefore, it is important to design and implement an appropriate intervention to improve the physical activity level, exercise self-efficacy, and cardiovascular risk factors in CHD patients in Sri Lanka. This study aims to develop and examine a culturally specific motivated, action-based intervention for improving physical activity level, exercise self-efficacy, and cardiovascular risk factors of CHD patients in Sri Lanka.

The participants will be patients who admitted to the coronary care unit (CCU) and medical wards of the Teaching Hospital Batticaloa, Sri Lanka with CHD for the first time confirmed by electrocardiogram with aged 18 years or above, able to reads and speak Tamil, able to attend clinic follow-up, obtain a medical clearance from a cardiologist to perform the exercise and, able to understand and give informed consent. The medical records of the CHD patients will be reviewed to screen for their eligibility. In addition, the cardiologist of the participants will be consulted for their suitability to perform the exercise of the intervention.

The purpose of the study, the data collection procedures, the potential risk and benefits, the maintenance of confidentiality, and the voluntary basis of participation will be clearly explained to the participants, and informed written consent will be obtained before data collection. Ethical approval was obtained from The Joint Chinese University of Hong Kong - New Territories East Cluster Clinical Research Ethics Committee and Ethics Review Committee, Faculty of Health Care-sciences, Eastern University, Sri Lanka.

The Statistical Package for Social Science version 22.0 software (SPSS 22.0) will be used to analyze the data and the p-value less than 0.5 will be considered as significant.

This study will provide evidence on the effectiveness of a motivated, action-based intervention on the physical activity level, cardiovascular risk factors, and exercise self-efficacy of CHD patients in Sri Lanka. Findings from this study could be useful to promote healthy lifestyle behaviors in CHD patients in a low-resource setting. Furthermore, this study will provide information on which level this intervention could be applied and possible constraints that hinder the outcomes of the results.

ELIGIBILITY:
Inclusion Criteria:

The eligibilities of participants are;

* Adults aged 18 years or above;
* Patients admitted to hospital with CHD for the first time confirmed by electrocardiogram;
* Patients able to reads and speak Tamil;
* Patients able to attend clinic follow-up, and obtain a medical clearance from a cardiologist to perform the exercise. The medical records of the CHD patients will be reviewed to screen for their eligibility. In addition, the cardiologist and physiotherapist at the study hospital will be consulted for confirming the suitability of the participants to perform the exercise of the intervention.

Exclusion Criteria:

The exclusion criteria are;

* Patients with absolute and relative contradictions to perform the exercise or at high risk for exercise, namely rest ejection fraction less than 40%, history of cardiac arrest, complex dysrhythmias at rest or during exercise testing or recovery, complicated myocardial infarction, high level of silent ischemia during exercise testing or recovery, presence of abnormal hemodynamics with exercise testing or recovery and presence of angina or other significant symptoms according to the American College of Sports Medicine (ACSM) guideline and American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR) guideline (American College of Sports Medicine [ACSM], 2014);
* Patients with any diagnosis of life-threatening conditions;
* Patients with the psychotic disease;
* Patients who unable to perform physical activity independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity level | Change from baseline physical activity level at 3 months.
  The validated Tamil version of International Physical Activity Questionnaire Short Form (IPAQ-SF) will be used to assess the self-reported time spent in walking, moderate and vigorous-intensity activities, and sitting in this study

SECONDARY OUTCOMES:
Change in cardiac exercise self-efficacy score | Change from baseline cardiac exercise self-efficacy score at 3 months.
  It will be measured using validated Tamil version of Cardiac Exercise Self-Efficacy Instrument (CESEI-T).The CESEI-T is a 16-item instrument to assess the individual's confidence to perform physical exercise in cardiac patients. Each item is rated on a five-point Likert scale from 1 (very little confidence) to 5 (quite a lot of confidence). Participants will be asked to rate their confidence level in performing exercise in various situations such as "fitting exercise into a busy day," "exercising without getting chest pain," "taking own heart rate before and after exercise," and "enduring light exercise". The CESEI-T score range from 16-80 and a higher score indicates that a high level of self-efficacy in performing the exercise.
Change in Body mass index (BMI) | Change from baseline body mass index at 3 months.
  All anthropometric measurements will be performed by a trained research assistant who will be blinded to the group allocation of participants. The weight will be measured with a calibrated mechanical personal scale. Participants will be weighed wearing light clothes, without shoes, and an empty bladder. The height will be measured in a standing position by using a plastic flexible tape (without shoes) and BMI will be calculated as weight in kilograms divided by height squared in meters (kg/m2).
Change in both Systolic Blood Pressure and Diastolic Blood Pressure | Change from baseline Systolic Blood Pressure and Diastolic Blood Pressure at 3 months.
  Blood pressure in a sitting position will be measured using a mercury sphygmomanometer (Dekamevit model Code: AC0125). Participants will be asked to rest for 15 minutes and no caffeinated food or drink 30 minutes before the blood pressure measurement.
Change in Fasting Blood Glucose (FBG) level | Change from baseline Fasting Blood Glucose level at 3 months.
  The participants' FBG level will be obtained from their clinical records.
Change in Waist hip ratio (WHR) | Change from baseline Waist hip ratio at 3 months.
  Waist circumference (WC) will be measured using a non-stretchable measuring tape at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest to the nearest 1cm, at end of the normal expiration. Hip circumference (HC) will be measured at the widest level over the grater trochanters using plastic flexible tape to the nearest 0.1 cm. WHR will be estimated as waist measurement (cm) divided by hip measurement (cm).
Change in total cholesterol level | Change from baseline total cholesterol level at 3 months.
  The participants' total cholesterol level will be obtained from their clinical records.
Change in high-density lipoprotein level | Change from baseline high-density lipoprotein level at 3 months.
  The participants' high-density lipoprotein level will be obtained from their clinical records.
Change in low-density lipoprotein level | Change from baseline low-density lipoprotein level at 3 months.
  The participants' low-density lipoprotein level will be obtained from their clinical records.
Change in triglyceride level | Change from baseline triglyceride level at 3 months.
  The participants' triglyceride level will be obtained from their clinical records.
Change in total cholesterol high-density lipoprotein ratio | Change from baseline total cholesterol high-density lipoprotein ratio at 3 months.
  The participants' total cholesterol high-density lipoprotein ratio will be obtained from their clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yu Cheng, PhD, Study Chair — Chinese University of Hong Kong
Locations (1):
- Teaching Hospital Batticaloa, Sri Lanka, Batticaloa, Eastern Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared with other researchers.

REFERENCES:
- [Derived] Karthijekan K, Cheng HY. Effectiveness of a motivated, action-based intervention on improving physical activity level, exercise self-efficacy and cardiovascular risk factors of patients with coronary heart disease in Sri Lanka: A randomized controlled trial protocol. PLoS One. 2022 Jul 5;17(7):e0270800. doi: 10.1371/journal.pone.0270800. eCollection 2022. PMID 35788765